CLINICAL TRIAL: NCT01978912
Title: Open-Label, Non-controlled, Single Ascending Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Exploratory Efficacy of KTP-001 in Subjects With Lumbar Disc Herniation
Brief Title: A Study to Evaluate Safety and Exploratory Efficacy of KTP-001 in Subjects With Lumbar Disc Herniation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Teijin America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KTP-001-CL-101
Record Dates: First submitted 2013-10-22; First posted 2013-11-08 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): one time 5 μg/disc dose of KTP-001 by intradiscal injection
  Interventions: Drug: KTP-001
- Cohort 2 (Experimental): one time 15 μg/disc dose of KTP-001 by intradiscal injection
  Interventions: Drug: KTP-001
- Cohort 3 (Experimental): one time 50 μg/disc dose of KTP-001 by intradiscal injection
  Interventions: Drug: KTP-001
- Cohort 4 (Experimental): one time 150 μg/disc dose of KTP-001 by intradiscal injection
  Interventions: Drug: KTP-001

INTERVENTIONS:
Drug: KTP-001 — KTP-001 is one time dose intradiscally.

SUMMARY:
The purpose of this study is to evaluate the safety and exploratory efficacy of KTP-001 in subjects with lumbar disc herniation.

DETAILED DESCRIPTION:
This study was a first-in-human, open-label, non-controlled single ascending dose study of KTP-001 in male and female subjects between the ages of 30 and 70 years with a single herniated lumbar disc. After obtaining informed consent, subjects were evaluated during a screening period of no more than 3 weeks (21 days). This study was conducted in 10 centers in the US.

Subjects that met all screening requirements and inclusion criteria and none of the exclusion criteria were enrolled into the study. Overall, 24 subjects were enrolled and treated: 6 subjects in each cohort. Cohort 1 received a 5 μg/disc dose of KTP-001 by intradiscal injection. Following administration of study drug, subjects were confined to the study center for 24 hours to collect data for safety and efficacy measures and collect blood samples for safety, PK evaluation, exploratory PD and anti-KTP-001 antibody and then returned for further assessments at various intervals from weeks 1 through to month 24.

After all subjects in Cohort 1 had received study drug, safety measures were evaluated by a Data and Safety Monitoring Board (DSMB) to determine whether to escalate KTP-001 administration to the next dose level. If appropriate, Cohort 2 subjects received 15 μg/disc of KTP-001, Cohort 3 subjects received 50 μg/disc of KTP-001, and Cohort 4 subjects received 150 μg/disc of KTP-001 by intradiscal injection. All safety, PK, and exploratory efficacy assessments were performed for the subjects in the subsequent cohorts as were performed for Cohort 1.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had a single contained or noncontained (extruded) lumbar disc herniation (L3-L4, L4-L5 or L5-S1) diagnosed by clinical symptoms and/or physical findings and confirmed by MRI.
* Subject has leg pain with a documented positive straight leg raise (SLR) test or femoral stretch test (FST).
* Subject has experiences herniated disc symptoms for at least 6 weeks prior to the study without relief with pain medications and other therapies.
* Subject has a BMI of 18 to 35 kg/m2

Exclusion Criteria:

* Subject has a sequestered lumbar disc herniation or intrathecal herniation confirmed by MRI
* Subject has two or more symptomatic lumbar disc herniations
* Previous intradiscal therapeutic intervention or has had any lumbar surgery
* Presence of lumbar spine disease and/or deformity other than a lumbar disc herniation
* Active smoker or is unable to abstain from tobacco use for 2 weeks prior to study injection
* Subject has a history or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - HOPE Research Institute, LLC, Phoenix, Arizona
  - CORE Orthopaedic Medical Center, Encinitas, California
  - California Spine Diagnostic, San Francisco, California
  - Compass Research, LLC, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Chicago Anesthesia Pain Specialists, Chicago, Illinois
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - William Beaumont Hospital, Royal Oak, Michigan

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 KTP-001 5 μg/Disc; Cohort 2 KTP-001 15 μg/Disc; Cohort 3 KTP-001 50 μg/Disc; Cohort 4 KTP-001 150 μg/Disc: KTP-001: KTP-001 is one time dose intradiscally.
Period: Overall Study
Arm/Group | Cohort 1 KTP-001 5 μg/Disc | Cohort 2 KTP-001 15 μg/Disc | Cohort 3 KTP-001 50 μg/Disc | Cohort 4 KTP-001 150 μg/Disc
Started | 6 | 6 | 6 | 6
Completed | 3 | 3 | 3 | 3
Not Completed | 3 | 3 | 3 | 3
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 2
Not completed — Lumbar Surgery | 1 | 0 | 1 | 0
Not completed — Intradiscal Steroid Injection | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 KTP-001 5 μg/Disc | Cohort 2 KTP-001 15 μg/Disc | Cohort 3 KTP-001 50 μg/Disc | Cohort 4 KTP-001 150 μg/Disc | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (3.33) | 49.0 (8.90) | 52.2 (13.23) | 47.0 (9.49) | 46.1 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 3 | 3 | 14
  Male | 1 | 3 | 3 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 0 | 4
  Not Hispanic or Latino | 4 | 5 | 5 | 6 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 2 | 3
  White | 5 | 6 | 6 | 4 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety Assessed by Adverse Events, Magnetic Resonance Imaging (MRI), X-ray Imaging, Physical Examination, Neurologic Examination and Vital Signs
Description: Any clinically significant changes were recorded as adverse events. They are described in the adverse events section of the results.
  AEs related to MRI, X-ray Imaging, Physical examination, and Neurologic examination are considered as adverse events of special interest (AESI). A treatment-emergent AE (TEAE) was defined as an AE that was not present prior to treatment with study drug, but appeared following treatment or was present at treatment initiation but worsened in severity during treatment.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 KTP-001 5 μg/Disc | Cohort 2 KTP-001 15 μg/Disc | Cohort 3 KTP-001 50 μg/Disc | Cohort 4 KTP-001 150 μg/Disc
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Participants with any AEs | 6 | 6 | 6 | 5
  Participants with any TEAEs | 6 | 6 | 6 | 5
  Participants with any serious TEAEs | 1 | 2 | 1 | 0
  Participants with any AESIs | 4 | 4 | 3 | 2
  TEAEs leading to study discontinuation | 0 | 1 | 0 | 0

2. Primary Outcome: Number of Participants With Change in 12-lead Electrocardiogram (ECG) and Clinical Laboratory Tests (CLT)
Description: Assessment of the number of participants with change in 12-lead ECG and CLT were assessed from baseline, 24 hours and 13 weeks.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 KTP-001 5 μg/Disc | Cohort 2 KTP-001 15 μg/Disc | Cohort 3 KTP-001 50 μg/Disc | Cohort 4 KTP-001 150 μg/Disc
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Participants with abnormal changes in ECG | 0 | 0 | 0 | 0
  Participants without abnormal changes in ECG | 6 | 6 | 6 | 6
  Participants with abnormal CLT | 0 | 0 | 0 | 0
  Participants without abnormal CL | 6 | 6 | 6 | 6

3. Secondary Outcome: Number of Participants Serum Concentrations of KTP-001 Below the Limit of Quantification (BLQ)
Description: The serum concentrations of KTP-001 were below the limit of quantification (BLQ) (<100 ng/mL) at all time points in all participants
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 KTP-001 5 μg/Disc | Cohort 2 KTP-001 15 μg/Disc | Cohort 3 KTP-001 50 μg/Disc | Cohort 4 KTP-001 150 μg/Disc
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  BLQ during the study up to 13 weeks | 6 | 6 | 6 | 6
  Not BLQ during the study up to 13 weeks | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Anti-KTP-001 Antibody
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 KTP-001 5 μg/Disc | Cohort 2 KTP-001 15 μg/Disc | Cohort 3 KTP-001 50 μg/Disc | Cohort 4 KTP-001 150 μg/Disc
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Negative during the study up to 13 weeks | 6 | 6 | 6 | 6
  Positive during the study up to 13 weeks | 0 | 0 | 0 | 0

5. Other Pre Specified Outcome: Changes in Lower Back Pain or Leg Pain Assessed by 11-point Numerical Rating Scale
Description: Lower back and leg pain were assessed using an 11-point numerical rating scale (0 = "no pain" and 10 = "worst possible pain").
  The endpoint was mean change from baseline at 6 and 13 weeks post-dose; with a negative number suggesting an improvement in pain while a positive number suggests a worsening in pain.
Time Frame: Baseline, 6 weeks and 13 weeks post-dose
Population: The Full Analysis Set (FAS) was used which consists of any subject who was enrolled into the study, received study drug, and had at least 1 efficacy evaluation after receiving study drug. In some cohorts, number of subjects are below 6 participants due to discontinuation and/or data missing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 KTP-001 5 μg/Disc | Cohort 2 KTP-001 15 μg/Disc | Cohort 3 KTP-001 50 μg/Disc | Cohort 4 KTP-001 150 μg/Disc
Number analyzed (Participants) | 6 | 6 | 6 | 6
score on a scale
  Change in Current Low Back Pain at Week 6: number analyzed (Participants) | 5 | 6 | 5 | 5
  Change in Current Low Back Pain at Week 6 | -3.6 (2.97) | -4.0 (2.28) | -3.2 (3.90) | -3.8 (1.79)
  Change in Current Low Back Pain at Week 13: number analyzed (Participants) | 5 | 6 | 6 | 5
  Change in Current Low Back Pain at Week 13 | -2.4 (2.61) | -3.7 (3.01) | -2.3 (4.18) | -2.8 (2.28)
  Change in Low Back Average Daily Pain at Week 6: number analyzed (Participants) | 5 | 6 | 5 | 5
  Change in Low Back Average Daily Pain at Week 6 | -3.64 (3.587) | -3.97 (2.448) | -3.36 (2.674) | -3.84 (2.551)
  Change in Low Back Average Daily Pain at Week 13: number analyzed (Participants) | 6 | 5 | 6 | 4
  Change in Low Back Average Daily Pain at Week 13 | -3.27 (2.919) | -4.36 (2.787) | -2.17 (3.572) | -4.30 (1.669)
  Change in Low Back Worst Daily Pain at Week 6: number analyzed (Participants) | 5 | 6 | 5 | 5
  Change in Low Back Worst Daily Pain at Week 6 | -3.72 (3.984) | -4.27 (3.066) | -3.64 (3.018) | -3.88 (2.488)
  Change in Low Back Worst Daily Pain at Week 13: number analyzed (Participants) | 6 | 5 | 6 | 4
  Change in Low Back Worst Daily Pain at Week 13 | -2.90 (2.928) | -4.96 (3.303) | -2.43 (3.829) | -2.90 (1.089)
  Change in Current Leg Pain at Week 6: number analyzed (Participants) | 5 | 6 | 5 | 5
  Change in Current Leg Pain at Week 6 | -2.8 (3.42) | -4.2 (1.83) | -4.2 (3.96) | -4.4 (2.70)
  Change in Current Leg Pain at Week 13: number analyzed (Participants) | 5 | 6 | 6 | 5
  Change in Current Leg Pain at Week 13 | -3.4 (3.05) | -5.2 (1.83) | -3.8 (3.87) | -4.4 (3.13)
  Change in Leg Average Daily Pain at Week 6: number analyzed (Participants) | 5 | 6 | 5 | 5
  Change in Leg Average Daily Pain at Week 6 | -2.66 (3.669) | -4.83 (1.515) | -3.76 (2.985) | -4.00 (3.476)
  Change in Leg Average Daily Pain at Week13: number analyzed (Participants) | 6 | 5 | 6 | 4
  Change in Leg Average Daily Pain at Week13 | -2.63 (3.053) | -5.28 (1.145) | -4.20 (2.647) | -5.70 (1.669)
  Change in Leg Worst Daily Pain at Week 6: number analyzed (Participants) | 5 | 6 | 5 | 5
  Change in Leg Worst Daily Pain at Week 6 | -2.34 (3.449) | -4.93 (2.355) | -4.12 (3.239) | -3.72 (3.294)
  Change in Leg Worst Daily Pain at Week13: number analyzed (Participants) | 6 | 5 | 6 | 4
  Change in Leg Worst Daily Pain at Week13 | -2.30 (3.074) | -5.60 (2.159) | -4.23 (2.986) | -5.40 (1.275)

6. Other Pre Specified Outcome: Number of Participants With Changes to Spinal Flexion and Tension Using the Straight-Leg Rising and/or Femoral Stretch Test
Description: The changes to spinal flexion and tension were assessed using Straight-Leg Rising (SLR) and Femoral Stretch (FS) tests which are on a scale of no change, positive to negative or negative to positive and where a positive result for SLR may indicate between 30 and 70 degrees, where a positive result for FS may indicate pain in the anterior thigh of the test leg and the elicited pain.
Time Frame: Baseline, 6 weeks and 13 weeks post-dose
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 KTP-001 5 μg/Disc | Cohort 2 KTP-001 15 μg/Disc | Cohort 3 KTP-001 50 μg/Disc | Cohort 4 KTP-001 150 μg/Disc
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Straight-Leg Raising Test at Week 6: Positive to Negative | 3 | 6 | 4 | 4
  Straight-Leg Raising Test at Week 6: Negative to Positive | 0 | 0 | 0 | 0
  Straight-Leg Raising Test at Week 6: No change | 2 | 0 | 1 | 1
  Straight-Leg Raising Test at Week 6: Missing | 1 | 0 | 1 | 1
  Straight-Leg Raising Test at Week 13: Positive to Negative | 4 | 6 | 4 | 4
  Straight-Leg Raising Test at Week 13: Negative to Positive | 0 | 0 | 0 | 0
  Straight-Leg Raising Test at Week 13: No change | 2 | 0 | 2 | 1
  Straight-Leg Raising Test at Week 13: Missing | 0 | 0 | 0 | 1
  Femoral Stretch Test at Week 6: Positive to Negative | 0 | 0 | 1 | 0
  Femoral Stretch Test at Week 6: Negative to Positive | 0 | 0 | 0 | 0
  Femoral Stretch Test at Week 6: No change | 5 | 6 | 4 | 5
  Femoral Stretch Test at Week 6: Missing | 1 | 0 | 1 | 1
  Femoral Stretch Test at Week 13: Positive to Negative | 1 | 0 | 2 | 0
  Femoral Stretch Test at Week 13: Negative to Positive | 0 | 0 | 0 | 0
  Femoral Stretch Test at Week 13: No change | 5 | 6 | 4 | 5
  Femoral Stretch Test at Week 13: Missing | 0 | 0 | 0 | 1

7. Other Pre Specified Outcome: Number of Participants With Changes in the Oswestry Disability Index
Description: The Oswestry Disability Index (ODI) score is calculated as participant score divided by possible score multiplied by 100, where the following scores can be interpreted to indicate:
  0-20% = Minimal disability; 20-40% = Moderate disability; 40-60% = Severe disability; 60-80% = Crippled; 80-100% = Bed bound;
Time Frame: Baseline, 6 weeks and 13 weeks post-dose
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 KTP-001 5 μg/Disc | Cohort 2 KTP-001 15 μg/Disc | Cohort 3 KTP-001 50 μg/Disc | Cohort 4 KTP-001 150 μg/Disc
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Baseline: 0-20 Minimal Disability | 0 | 0 | 0 | 0
  Baseline: 20-40 Moderate Disability | 3 | 2 | 1 | 3
  Baseline: 40-60 Severe Disability | 2 | 3 | 4 | 1
  Baseline: 60-80 Crippled | 1 | 1 | 1 | 2
  Baseline: 80-100 Bedbound | 0 | 0 | 0 | 0
  Baseline: missing | 0 | 0 | 0 | 0
  Week 6: 0-20 Minimal Disability | 2 | 1 | 2 | 3
  Week 6: 20-40 Moderate Disability | 2 | 5 | 3 | 2
  Week 6: 40-60 Severe Disability | 0 | 0 | 0 | 0
  Week 6: 60-80 Crippled | 0 | 0 | 0 | 0
  Week 6: 80-100 Bedbound | 1 | 0 | 0 | 0
  Week 6: missing | 1 | 0 | 1 | 1
  Week 13: 0-20 Minimal Disability | 2 | 3 | 3 | 4
  Week 13: 20-40 Moderate Disability | 2 | 3 | 2 | 1
  Week 13: 40-60 Severe Disability | 1 | 0 | 1 | 0
  Week 13: 60-80 Crippled | 1 | 0 | 0 | 0
  Week 13: 80-100 Bedbound | 0 | 0 | 0 | 0
  Week 13: missing | 0 | 0 | 0 | 1

8. Other Pre Specified Outcome: Changes in Quality of Life as Assessed by Short Form-12 (SF-12)
Description: The endpoint was change from baseline at Week 6 and 13 hours post-dose. The Short Form-12 (SF-12) is a Quality of Life questionnaire which measures functional health and well-being from a participant's perspective across eight health domains. Each participant answers questions on a 5-point Likert scale, which rates responses according to how much the participant agrees or disagrees with a particular statement on their health and wellbeing, including vitality/physical functioning/bodily pain/general health perceptions/physical role functioning/emotional role functioning/social role functioning and mental health. Each scale is transformed into a 0-100 scale, assuming each question carries equal weight. Lower scores mean greater disability and higher scores mean less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: Baseline, 6 weeks and 13 weeks post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 KTP-001 5 μg/Disc | Cohort 2 KTP-001 15 μg/Disc | Cohort 3 KTP-001 50 μg/Disc | Cohort 4 KTP-001 150 μg/Disc
Number analyzed (Participants) | 6 | 6 | 6 | 6
score on a scale
  Change in Physical Functioning score at Week 6: number analyzed (Participants) | 5 | 6 | 5 | 5
  Change in Physical Functioning score at Week 6 | 0.400 (0.4183) | 0.333 (0.3028) | 0.400 (0.4183) | 0.200 (0.2092)
  Change in Physical Functioning score at Week 13: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change in Physical Functioning score at Week 13 | 0.208 (0.2458) | 0.500 (0.3162) | 0.333 (0.5401) | 0.250 (0.2500)
  Change in Role Physical score at Week 6: number analyzed (Participants) | 5 | 6 | 5 | 5
  Change in Role Physical score at Week 6 | 0.2500 (0.35355) | 0.2292 (0.27858) | 0.3000 (0.20917) | 0.2250 (0.31125)
  Change in Role Physical score at Week 13: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change in Role Physical score at Week 13 | 0.1667 (0.23274) | 0.2083 (0.32275) | 0.3333 (0.41583) | 0.3750 (0.15309)
  Change in Bodily Pain score at Week 6: number analyzed (Participants) | 5 | 6 | 5 | 5
  Change in Bodily Pain score at Week 6 | -0.100 (0.3791) | -0.417 (0.2041) | -0.300 (0.2739) | -0.350 (0.1369)
  Change in Bodily Pain score at Week 13: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change in Bodily Pain score at Week 13 | -0.167 (0.3764) | -0.417 (0.2041) | -0.333 (0.3028) | -0.400 (0.2850)
  Change in General Health score at Week 6: number analyzed (Participants) | 5 | 6 | 5 | 5
  Change in General Health score at Week 6 | 0.000 (0.0000) | 0.042 (0.1021) | -0.100 (0.1369) | -0.150 (0.1369)
  Change in General Health score at Week 13: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change in General Health score at Week 13 | 0.000 (0.0000) | -0.042 (0.1021) | -0.167 (0.1291) | -0.100 (0.1369)
  Change in Vitality score at Week 6: number analyzed (Participants) | 5 | 6 | 5 | 5
  Change in Vitality score at Week 6 | -0.100 (0.2236) | -0.167 (0.1291) | 0.050 (0.2092) | -0.250 (0.2500)
  Change in Vitality score at Week 13: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change in Vitality score at Week 13 | 0.000 (0.3162) | -0.125 (0.1369) | -0.042 (0.2923) | -0.200 (0.2739)
  Change in Social Functioning score at Week 6: number analyzed (Participants) | 5 | 6 | 5 | 5
  Change in Social Functioning score at Week 6 | 0.100 (0.2850) | 0.292 (0.2923) | 0.250 (0.2500) | 0.300 (0.2092)
  Change in Social Functioning score at Week 13: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change in Social Functioning score at Week 13 | 0.125 (0.2092) | 0.333 (0.3028) | 0.333 (0.3764) | 0.400 (0.2850)
  Change in Role Emotional score at Week 6: number analyzed (Participants) | 5 | 6 | 5 | 5
  Change in Role Emotional score at Week 6 | 0.1000 (0.34686) | 0.2292 (0.25516) | 0.2500 (0.19764) | 0.1750 (0.31375)
  Change in Role Emotional score at Week 13: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change in Role Emotional score at Week 13 | 0.1875 (0.27099) | 0.3542 (0.30017) | 0.2083 (0.20412) | 0.2750 (0.32355)
  Change in Mental Health score at Week 6: number analyzed (Participants) | 5 | 6 | 5 | 5
  Change in Mental Health score at Week 6 | 0.0000 (0.08839) | 0.0625 (0.06847) | 0.0250 (0.13693) | -0.0500 (0.22707)
  Change in Mental Health score at Week 13: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change in Mental Health score at Week 13 | -0.0417 (0.06455) | 0.1667 (0.21890) | 0.0208 (0.14613) | 0.0250 (0.16298)

9. Other Pre Specified Outcome: Patient Global Impression of Change (PGI-C)
Description: The Patient Global Impression Change PGI-C scale was used where the scale ranges are from 1 (no change or condition has got worse) to 7 (a great deal better, and a considerable improvement). The endpoint was the value at 6 and 13 weeks post-dose.
Time Frame: Baseline, 6 weeks and 13 weeks post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 KTP-001 5 μg/Disc | Cohort 2 KTP-001 15 μg/Disc | Cohort 3 KTP-001 50 μg/Disc | Cohort 4 KTP-001 150 μg/Disc
Number analyzed (Participants) | 6 | 6 | 6 | 6
score on a scale
  Week 6: number analyzed (Participants) | 5 | 6 | 5 | 5
  Week 6 | 4.4 (3.78) | 2.3 (1.37) | 3.2 (3.27) | 2.2 (1.64)
  Week 13: number analyzed (Participants) | 6 | 6 | 6 | 5
  Week 13 | 4.7 (2.34) | 2.2 (1.17) | 3.3 (3.27) | 2.8 (2.39)

10. Other Pre Specified Outcome: Changes in Serum Concentrations of Keratan Sulfate
Description: The endpoint was change from baseline at 6 and 24 hours post-dose, and at the 1-, 2-, 4-, 6-, and 13-week follow-up visits or early termination visit.
Time Frame: Baseline, 6 and 24 hours and 1, 2, 4, 6 weeks and 13 weeks post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 KTP-001 5 μg/Disc | Cohort 2 KTP-001 15 μg/Disc | Cohort 3 KTP-001 50 μg/Disc | Cohort 4 KTP-001 150 μg/Disc
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/ml
  6 hours | -93.7 (59.22) | -84.7 (47.24) | -37.3 (42.28) | -24.8 (49.68)
  24 hours | -39.2 (87.90) | -73.2 (34.59) | 35.2 (72.37) | 141.8 (262.07)
  Week 1 | 77.3 (30.66) | 47.2 (47.31) | 117.7 (41.31) | 297.3 (144.99)
  Week 2: number analyzed (Participants) | 6 | 6 | 5 | 6
  Week 2 | 47.0 (62.77) | 22.2 (81.96) | 102.0 (69.13) | 173.2 (120.44)
  Week 4: number analyzed (Participants) | 6 | 6 | 5 | 6
  Week 4 | -6.2 (45.44) | -36.7 (66.22) | 87.2 (49.60) | 26.8 (79.08)
  Week 6: number analyzed (Participants) | 5 | 6 | 5 | 5
  Week 6 | 1.4 (74.31) | -41.7 (69.84) | 64.0 (61.46) | 11.0 (81.86)
  Week 13: number analyzed (Participants) | 6 | 6 | 6 | 5
  Week 13 | -7.5 (127.30) | -39.2 (63.90) | 55.8 (83.71) | -13.6 (43.64)

ADVERSE EVENTS:
Time Frame: 24 month
Arm/Group | Cohort 1 KTP-001 5 μg/Disc | Cohort 2 KTP-001 15 μg/Disc | Cohort 3 KTP-001 50 μg/Disc | Cohort 4 KTP-001 150 μg/Disc
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 KTP-001 5 μg/Disc (N=6) | Cohort 2 KTP-001 15 μg/Disc (N=6) | Cohort 3 KTP-001 50 μg/Disc (N=6) | Cohort 4 KTP-001 150 μg/Disc (N=6)
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 KTP-001 5 μg/Disc (N=6) | Cohort 2 KTP-001 15 μg/Disc (N=6) | Cohort 3 KTP-001 50 μg/Disc (N=6) | Cohort 4 KTP-001 150 μg/Disc (N=6)
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 3 | 1 | 3
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Radicular pain (Nervous system disorders) | 0 | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2015-10-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT01978912/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT01978912/SAP_001.pdf